CLINICAL TRIAL: NCT07006870
Title: Impact of Adding Virtual Reality Training to Balance Exercise Training Program on Balance, Postural Stability, Mobility and Quality of Life in Obese Patients, A Prospective Randomized Controlled Trial
Brief Title: Virtual Reality Training on Balance, Postural Stability, Mobility and Quality of Life in Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 005842
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Obesity/Therapy; Obesity (Body Mass Index >30 kg/m2)
Keywords: Virtual Reality Training; Balance; Postural Stability; Quality of Life; Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality Plus Balance exerciseTraining Group (Experimental): 30 patients will receive Virtual reality training in addition to balance exercise program. for 30 minutes, 3 days/ week for 8 weeks.
  Interventions: Other: Virtual Reality plus Balance Exercise Training; Other: Balance Exercise Training
- Balance Training Exercise Program (Active Comparator): 30 patients will receive balance exercise program. for 30 minutes, 3 days/ week for 8 weeks.
  Interventions: Other: Balance Exercise Training

INTERVENTIONS:
Other: Virtual Reality plus Balance Exercise Training — Virtual reality balance training will be completed using the BRU system's preloaded programs for postural training and rehabilitation. Rehabilitation exercises will include tasks performed standing with virtual reality headset on whereby the visual and vestibular systems will be stressed and will be customized according to the participant's needs and ability to tolerate the training stimulus. Postural training exercises will be used to develop limits of stability, with 3 exercises performed requiring participants to move their center of mass to collect rings/blocks through a course within a given amount of time. Each of the 3 postural training exercises contained 15 levels of varying difficulty. Sessions will be tailored to everyone, with progression of increasing the level of difficulty or time of exposure for each exercise. Participants at this group will be also participate in a Balance exercise training program for 40 min/3 times per week for 8 weeks.
  Arms: Virtual reality Plus Balance exerciseTraining Group
Other: Balance Exercise Training — Each session of balance exercises will be composed of three phases, including warm-up, balance training and cool down. The warm-up phase will involve gentle stretching for calf, hamstring, quadriceps, iliopsoas muscles, as well as anterior, posterior and lateral step-ups for 5-10 minutes. The active phase will be performed on a balance training for 20 minutes. It included heel and toe raises, one-legged stance for each extremity, shifting weight anteriorly, posteriorly, laterally and diagonally, step-ups, narrow walking, backward walking, sideward walking, stepping over obstacles, passing balls arranged on the training mat in a circle, and throwing and catching a ball on the training mat. A rest period of 1 minute will be given between each component. The program will be ended with 5-10 minutes of cool down. During the cool-down phase, patients will perform deep breathing exercises and static exercises for back extensors in a recumbent position.

SUMMARY:
The aim of this study will be to evaluate the effect of adding Virtual reality training to balance exercise program on improving Balance, Postural Stability, mobility and Quality of life in obese patients.

ELIGIBILITY:
Inclusion criteria:

1. Participants with 20 to 40 years old,
2. Participants with BMI of 30 to 39.9 kg/m2
3. Absence of neurological disorders i.e.: stroke, ataxia, or parkinsonism.

Exclusion criteria:

1. Participants with vestibular or vision problem.
2. Participants with Diabetes mellitus or cardiorespiratory disorders.
3. Participants with severe obesity BMI ≥40.
4. participants at regular physical therapy exercise training program at the last 3 months.
5. Participants who are unable to follow instructions due to personal or cognitive problems.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Single-Leg Stance Test | Eight weeks
  Single-Leg Stance Test on Firm and Foam Surfaces Participants were asked to stand on 1 leg with eyes open on firm and foam surfaces for as long as possible; the time in seconds was recorded using a stopwatch. Participants completed 3 trials on each leg, and a mean score was calculated for each leg. Rest was permitted between each trial. The test was terminated when (1) the raised foot touched the stance leg or the floor, (2) the participant hopped, and (3) the arm touched a support surface or the investigator. The dominant leg was indicated by the preferred foot when kicking a ball. This test has shown excellent test-retest reliability among healthy older adults, and predictive validity in older adults with Parkinson disease. A cutoff of <10 seconds has discriminated between fallers and non-fallers with Parkinson disease

SECONDARY OUTCOMES:
Stability Assessment | Eight weeks.
  The Biodex Balance System (Biodex Medical System, Inc., Shirley, NY, USA) will be used to measure anteroposterior, mediolateral, and overall stability indices. Postural balance assessment will evaluate the participant's ability to regulate the platform's tilt angle, with deviations from the centre using standard deviation instead of the mean. Each test will last 20 seconds, with a 10-minute rest between three trials. The Biodex Balance System is reported to have high reliability
Timed-Up-and-Go Test | Eight weeks.
  The TUG test involved participants' getting up from a chair, walking 3 meters at a comfortable speed, turning around, walking back to the chair, and sitting down.45 The time in seconds was recorded between when the examiner verbalized "go" and when the participants back touched the backrest of the chair. The average of the 2 experimental trials was used in the analysis. The test has shown high inter- and intrarater reliability,53 as well as discriminative validity in community dwelling and institutionalized older adults.5 A clinical cutoff of ≤12 seconds has been a recognized threshold for normal TUG performance in community-dwelling older adults
The Short Form-36 (SF-36) Questionnaire | Eight weeks
  It will be used to evaluate quality of life. This instrument assesses eight domains: general health, mental health, physical functioning, role physical, role emotional, body pain, social functioning, and vitality. Scores for each domain range from 0 to 100, with 0 representing the worst and 100 the best quality of life. The SF-36 primarily evaluates physical and mental aspects and has demonstrated validity and reliability in burn survivors

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Access Criteria: After 6 months of publication

REFERENCES:
- [Result] Sadeghi H, Jehu DA, Daneshjoo A, Shakoor E, Razeghi M, Amani A, Hakim MN, Yusof A. Effects of 8 Weeks of Balance Training, Virtual Reality Training, and Combined Exercise on Lower Limb Muscle Strength, Balance, and Functional Mobility Among Older Men: A Randomized Controlled Trial. Sports Health. 2021 Nov-Dec;13(6):606-612. doi: 10.1177/1941738120986803. Epub 2021 Feb 13. PMID 33583253
- [Result] Fang Q, Ghanouni P, Anderson SE, Touchett H, Shirley R, Fang F, Fang C. Effects of Exergaming on Balance of Healthy Older Adults: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Games Health J. 2020 Feb;9(1):11-23. doi: 10.1089/g4h.2019.0016. Epub 2019 Dec 3. PMID 31800322
- [Result] Anastasiadou D, Herrero P, Garcia-Royo P, Vazquez-De Sebastian J, Slater M, Spanlang B, Alvarez de la Campa E, Ciudin A, Comas M, Ramos-Quiroga JA, Lusilla-Palacios P. Assessing the Clinical Efficacy of a Virtual Reality Tool for the Treatment of Obesity: Randomized Controlled Trial. J Med Internet Res. 2024 Apr 5;26:e51558. doi: 10.2196/51558. PMID 38578667
- [Result] Greco G, Poli L, Gabriele M, Aidar FJ, Fischetti F, Patti A, Cataldi S. Effectiveness of a 5-week virtual reality versus traditional training on balance and flexibility in healthy adult females. Sport Sciences for Health. 2025 Mar;21(1):289-300.